CLINICAL TRIAL: NCT00461565
Title: A Double Blind, Randomized, Placebo Controlled, Two Part, Two Session Balanced, Crossover Study to Evaluate Visual Changes in Healthy Male Subjects Aged 18 - 55 Years After Receiving: 1. at Least 15 Doses of 20 mg Vardenafil, Compared to Placebo and 2. Two Doses of Sildenafil, 200 mg Compared to Placebo
Brief Title: FDA Phase IV - Commitment - Retinal Function Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11337; VAR 102 162 (Other: Company internal)
Record Dates: First submitted 2007-04-17; First posted 2007-04-18 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: Safety
Keywords: Retina; PDE-5; Levitra; Viagra; Normal healthy volunteers for evaluation of retinal function
MeSH Terms: interventions — Sildenafil Citrate; Vardenafil Dihydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Part A1 (Active Comparator)
  Interventions: Drug: Sildenafil
- Part A2 (Placebo Comparator)
  Interventions: Drug: Placebo
- Part B1 (Experimental)
  Interventions: Drug: Vardenafil (Levitra, BAY38-9456)
- Part B2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sildenafil — A1) Two dosis of 200 mg Sildenafil orally. Patients receive either A1) or A2) in cross over design with either B1) or B2).
  Arms: Part A1
Drug: Placebo — A2) Matching Placebo orally. Patients receive either A1) or A2) in cross over design with either B1) or B2).
  Arms: Part A2
Drug: Vardenafil (Levitra, BAY38-9456) — B1) At least 15 dosis of 20 mg Levitra orally. Patients receive either A1) or A2) in cross over design with either B1) or B2).
  Arms: Part B1
Drug: Placebo — B2) Matching Placebo orally. Patients receive either A1) or A2) in cross over design with either B1) or B2).
  Arms: Part B2

SUMMARY:
Vardenafil (Levitra) and Sildenafil (Viagra) are drugs that are marketed for use in patients with erectile dysfunction. The purpose of this study is to find out if there are any changes in the eye after taking at least 15 doses of Vardenafil and after two doses of Sildenafil. This is a double-blind study, which means that neither you nor the study doctor will know which treatment you are receiving. If you qualify for the study, you will receive:- Vardenafil 20 mg twice per week (Monday and Thursday) for a maximum of 8 weeks. There will be two times when this occurs during the study.- Sildenafil 200 mg/day for two days. There will be two times when this occurs during the study. - Placebo (a pill that looks like vardenafil or sildenafil but has no active ingredient).

ELIGIBILITY:
Inclusion Criteria:- Healthy adult male subjects between 18 and 55 years of age, inclusive, at screening- Body mass index (BMI) 19 to 34 kg/m2- Negative for HIV, Hepatitis B and Hepatitis C at screening Exclusion Criteria:- Any unstable medical, psychiatric, or substance abuse disorder- History of moderate or severe hepatic impairment- Creatinine clearance- A resting systolic blood pressure of < 100 mm Hg or > 170 mm Hg or a resting diastolic blood pressure > 110 mm Hg- Blindness, color blindness or vision in either eye judged as abnormal by the investigator- History of trauma or surgery to either eye, of retinitis pigmentosa, of diabetes or current diabetes, of epilepsy or of seizure disorders- Symptomatic hypotension within 6 months of start of study- History of sickle cell anemia or sickle cell trait or bleeding disorder- Significant active peptic ulceration or other gastrointestinal disorder such as colitis or Crohn's Disease- Use of alpha blockers, nitrates, ritonavir, indinavir, ketoconazole, itraconazole, or erythromycin, ciprofloxacin, tadalafil, isotretinoin, ibuprofen, unoprostone isopropyl, Lily-of-the-Valley, Strophanthus, ranitidine and sildenafil

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2005-02; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
The change from baseline in Fansworth Munsell (FM) 100 test total error score (TES) in both the left and right eyes for vardenafil treated subjects as compared to placebo | 8 weeks

SECONDARY OUTCOMES:
The change from baseline in Electroretinogram (ERG) as measured by amplitude and implicit time of b wave in both the left and right eyes for vardenafil treated subjects as compared to placebo | 8 weeks
Change in the FM-100 total error score from baseline at approximately 6 hours and 24 hours post dose | 8 weeks
Safety and tolerability of 20 mg vardenafil after at least 15 oral doses of 20 mg vardenafil or placebo (dosed over approximately 8 weeks) | 8 weeks
ERG and FM-100 total error score from baseline at approximately 2 hours following one dose of sildenafil 200 mg | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer